CLINICAL TRIAL: NCT04827992
Title: Evaluation of Medical Cannabis and Prescription Opioid Taper Support for Reduction of Pain and Opioid Dose in Patients With Chronic Non-Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Cambridge Health Alliance (Other); MaineHealth (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jodi Gilman, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P000871; R01DA051540 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use; Pain; Marijuana Use
Keywords: Opioid; Marijuana; Pain; neurocognition; Dependence; Behavioral treatment
MeSH Terms: conditions — Pain; Marijuana Use; Marijuana Abuse | interventions — Medical Marijuana; nabiximols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Marijuana + Prescription Opioid Taper Support (POTS) behavioral treatment (Experimental): This group can begin using medical marijuana immediately and will participate in the POTS treatment groups.
  Interventions: Drug: Medical Marijuana; Behavioral: Prescription Opioid Taper Support (POTS)
- Prescription Opioid Taper Support (POTS) treatment alone (Active Comparator): This group must abstain from marijuana use and will participate in the POTS behavioral treatment alone.
  Interventions: Behavioral: Prescription Opioid Taper Support (POTS)

INTERVENTIONS:
Drug: Medical Marijuana — Patients in this group can choose what type, how much, and when to use medical marijuana to use.
  Other Names: Cannabis
  Arms: Medical Marijuana + Prescription Opioid Taper Support (POTS) behavioral treatment
Behavioral: Prescription Opioid Taper Support (POTS) — Prescription Opioid Taper Support (POTS), a manualized behavioral prescription opioid taper support intervention developed by consultant, will be offered weekly to all participants to support behavioral self-management of pain and structured, voluntary taper of COT dose.

SUMMARY:
This study will use a randomized controlled design to test whether medical marijuana use by adults on high-dose chronic opioid therapy (COT) for chronic non-cancer pain is associated with reduced opioid dose and improved pain intensity and interference when added to a 24-week behavioral intervention (POTS).

DETAILED DESCRIPTION:
This trial is a randomized, six-month study of medical marijuana (MM) on opioid use that will: (1) evaluate whether adults with chronic, non-cancer pain on COT assigned to MM+POTS, compared with those assigned to WL+POTS, have greater reduction in opioid dose and/or pain intensity and interference, (2) assess whether participants assigned to MM+POTS, compared with those assigned to WL+POTS, have improved quality of life, depression, and anxiety; and reduced self-reported opioid dose, (3) evaluate whether those assigned to MM+POTS develop symptoms of CUD and have a reduced number of OUD symptoms over the 24-week intervention, as well as at the 12-month time point.

Participants will be randomly assigned to either an active MM arm (n = 60), or to a waitlist control arm (WLC) (n = 60). Participants will be assessed at baseline, every 4 weeks for 6 months, and at a 12-month follow-up for opioid use, development of CUD, development or resolution of OUD, and neurocognitive performance. Urine collected will be assessed with quantitative assays.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-75, inclusive.
2. Endorsing > 6 months of chronic, non-cancer pain.
3. On stable prescription opioid doses of 25 MME or greater for >90 days, verified by the Prescription Monitoring Program.
4. Either no prior use or current light cannabis use (weekly or less in the past 12 months).
5. Plans to use medical cannabis for pain to control pain and/or reduce opioid dose.
6. Competent and willing to provide written informed consent in English.
7. Potential participants of childbearing potential must not be pregnant at enrollment. They will be asked to self-report pregnancy status and the start date of their most recent menstrual period and agree to use effective contraception: abstinence; hormonal contraception; intra-uterine device, sterilization; or double barrier contraception, during the study.

Exclusion Criteria:

1. Current cannabis use (including inhaled or ingested CBD products) of greater than weekly on average in the past 12 months, assessed via self-report (no more than 10 times in the past 90 days).
2. Current cannabis use disorder; current moderate to severe substance use disorder for any substance by structured interview, EXCEPT nicotine and opioids (OUD).
3. Current uncontrolled major medical illness, such as cancer, symptomatic hypothyroidism/hyperthyroidism or severe respiratory compromise.
4. Use of non-prescribed opioids, by self-report.
5. Dose change or initiation of medications with significant analgesic effects (e.g., tricyclic antidepressants, SSRIs, gabapentin, NSAIDs) in the past 4 weeks.
6. Concomitant medications will be discussed at each study visit, and any medications that may interact with cannabinoids (e.g., warfarin) will be discussed with a study clinician prior to enrollment or continued participation.
7. Actively suicidal and/or suicide attempt or psychiatric hospitalization in past year, or current suicidal ideation with specific plan or intent.
8. History of intellectual disability (e.g., Down's syndrome) or other severe developmental disorder or IQ < 70.
9. Current diagnosis of delirium, dementia, amnestic, or other cognitive disorder; current diagnosis of bipolar II disorder; lifetime diagnosis of bipolar I disorder, schizophrenia spectrum, or other psychotic disorder.
10. Surgery within the past month or planned during the next 6 months.
11. Pregnant or trying to get pregnant or breastfeeding.
12. In the opinion of the investigator or study physicians, not able to complete study procedures or safely participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Mean Difference in Prescription Monitoring Program verified opioid dose at baseline and week 24 | Week 24
  Median opioid dose verified by the Prescription Monitoring Program, in morphine milligram equivalents (MME) per day, over monthly interval preceding study visit.
Mean Difference in Pain, Enjoyment, General Activity (PEG) Scale Summed Score over post-baseline to week 24 interval | Every post-baseline day until week 24
  The Pain, Enjoyment, General Activity (PEG) scale will assess pain intensity and interference. The scale ranges from 0-30, with a higher score indicating greater pain intensity and interference. Collected daily by a self-reported online survey.

SECONDARY OUTCOMES:
Mean Difference in Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form Summed Score at weeks 4, 8, 12, 16, 20, 24 | Week 4, week 8, week 12, week 16, week 20, week 24
  Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form will assess changes in quality of life measures. The scale ranges from 14 - 70, with a lower score indicating greater dissatisfaction with life.
Mean Difference in PROMIS-29 Depression Subscale Summed Score at weeks 4, 8, 12, 16, 20, 24 | Week 4, week 8, week 12, week 16, week 20, week 24
  The 8-item depression subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 will be used to assess depression symptoms. The scale uses a t-score metric (mean of 50, SD of 10). Higher scores indicate worse depression.
Mean Difference in PROMIS-29 Anxiety Subscale Summed Score at weeks 4, 8, 12, 16, 20, 24 | Week 4, week 8, week 12, week 16, week 20, week 24
  The 7-item anxiety subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 will be used to assess anxiety symptoms. The scale uses a t-score metric (mean of 50, SD of 10). Higher scores indicate worse anxiety.
Mean Difference in Opioid Use Disorder Symptoms at weeks 4, 8, 12, 16, 20, 24 | Week 4, week 8, week 12, week 16, week 20, week 24
  The DSM-5 Opioid Use Disorder Checklist will evaluate symptoms of Opioid Use Disorder (number of symptoms). The scale ranges from 0 - 11, with a higher score indicating more severe Opioid Use Disorder.
Mean Difference in Cannabis Use Disorder Symptoms at weeks 12 and 24 | Week 12, Week 24
  The DSM-5 Cannabis Use Disorder Checklist will evaluate symptoms of Cannabis Use Disorder (number of symptoms). The scale ranges from 0 - 11, with a higher score indicating more severe Cannabis Use Disorder.
Mean Difference in Self-Reported Opioid Dose over post-baseline to week 24 interval | Every post-baseline day until week 24
  Self-reported opioid dose in morphine milligram equivalents (MME) per day.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Gilman, PhD, Principal Investigator — Massachusetts General Hospital; A. Eden Evins, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cambridge Health Alliance, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
All data, code, and materials used in the analyses can be provided by Jodi Gilman and Massachusetts General Hospital pending scientific review and a completed data use agreement/material transfer agreement beginning one year after publication of the results. Requests for all materials should be submitted to Jodi Gilman at jgilman1@mgh.harvard.edu.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available beginning one year after publication of the results.
Access Criteria: Data will be provided pending a scientific review and a completed data use agreement/material transfer agreement. Requests should be submitted to Jodi Gilman at jgilman1@mgh.harvard.edu

REFERENCES:
- [Background] Jashinski J, Grossman E, Quaye A, Cather C, Potter K, Schoenfeld DA, Evins AE, Gilman JM. Randomised, pragmatic, waitlist controlled trial of cannabis added to prescription opioid support on opioid dose reduction and pain in adults with chronic non-cancer pain: study protocol. BMJ Open. 2022 Jun 9;12(6):e064457. doi: 10.1136/bmjopen-2022-064457. PMID 35680252

DOCUMENTS (2):
  • Statistical Analysis Plan (2025-10-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT04827992/SAP_008.pdf
  • Informed Consent Form (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT04827992/ICF_007.pdf